CLINICAL TRIAL: NCT07002645
Title: The Effect of Web-Based Conflict Resolution Training Applied to Intensive Care Nurses on the Conflict Resolution Skills of Nurses
Brief Title: The Effect of Web-Based Conflict Resolution Training Applied to Intensive Care Nurses
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Özlem Canbolat, Gazi University, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: E-77082166-302.08.01-1131600
Record Dates: First submitted 2025-05-25; First posted 2025-06-03 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-05

CONDITIONS: Conflict Resolution; Intensive Care Nurses; Web-based Training
Keywords: conflict resolution; intensive care nurses; web-based training
MeSH Terms: conditions — Negotiating

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Application group (Experimental): After the purpose of the study and the method of application are explained to the intensive care nurses, the "Introductory Information Form", and Conflict Resolution Scale will be applied. Web-based conflict resolution training program will be applied to the intervention group for 2 week. The Conflict Resolution Scale will be repeated at the end of Web-based conflict resolution training program.The Web-Based Conflict Resolution Training Satisfaction Survey will be administered to the intervention group along with the post-test, which will question their satisfaction with the conflict resolution training program.
  Interventions: Other: Web-based conflict resolution training program
- Control Group (No Intervention): After explaining the purpose of the study and the way it was applied to patients in the control group, Introductory Information Form, and The Conflict Resolution Scale will be applied. No application will be made to the control group. The control group will be reapplied The Conflict Resolution Scale after two week the pretest.

INTERVENTIONS:
Other: Web-based conflict resolution training program — Researchers developed the content of the web-based conflict resolution training program. First, ten experts were consulted to check the program's clarity and suitability. Second, the program was revised and finalized according to the experts' feedback.
  A web page was obtained from the World Wide Web (www) by using hosting and domain services. Technical support and consultancy were received from a professional web design company during the implementation of the website. The content of the training program, for which expert opinions were obtained, was transferred to the web page. Web-based conflict resolution training program will be applied to the intervention group for 2 week.
  Arms: Application group

SUMMARY:
This study will be conducted in a randomized parallel controlled experimental study design to determine the effect of web-based conflict resolution training to be applied to intensive care nurses on the conflict resolution skills of nurses.

The study will be conducted with 46 nurse (23 intervention, 23 control groups) working in the Intensive Care Units of an University Hospital between May 2025 and September 2026.

Web-based conflict resolution training program will be applied to the intervention group for 2 week.No application will be made to the control group. The data collection tools in the study are the Identifier Information Form, Conflict Resolution Scale, and Satisfaction Survey for Web-Based Conflict Resolution Training.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Having worked in intensive care for at least six months
* Having access to the internet
* Able to use the internet
* Agree to participate in the study

Exclusion Criteria:

* Having a high school or associate degree,
* Having been temporarily assigned to an intensive care unit.
* Leaving the research voluntarily,
* Not completing the training sessions,
* Not participating in the activities in the Training Modules.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-05-25 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Conflict Resolution Scale | The Conflict Resolution Scale will be applied for pretest. The Conflict Resolution Scale will be reapplied after two week the pretest.
  Scores from the scale range from 55 to 220, and the higher the score, the higher conflict resolution skill level.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided